CLINICAL TRIAL: NCT05850897
Title: The Effect of Foot Massage Applied Before and After Cholecystectomy Surgery on Anxiety, Pain and Comfort Level
Brief Title: The Effect of Foot Massage on Anxiety, Pain and Comfort Level
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Nesibe Sultan ÇINAROĞLU, PhD Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: *SBU,SR,NSBÇ-44*
Record Dates: First submitted 2023-04-17; First posted 2023-05-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Pain; Anxiety
Keywords: Cholessystectomy; Foot massage; Comfort
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage Group (Experimental): Appropriate position is given to the patients. Thumb and finger movements, patting, rubbing and squeezing techniques are used in foot massage. During training, the active hand applies pressure, while the passive hand uses both hands to support the foot. The intervention begins with rubbing and warming the feet. The duration of the foot warming process is approximately 5 minutes, and after the foot warming maneuvers, the methods of moving the thumbs of both hands towards the soles of the feet and spinning the laundry are used. The inner and outer parts of the foot are patted in a balanced way. This caressing movement on both feet is done with these movements in a light and rhythmic way and the massage is completed. Data will be obtained with Patient Descriptive Information Form, Vital Signs Follow-up Form, Surgical Anxiety Scale for Adult Patients, Perianesthesia Comfort Scale, Numerical Pain Scale.
  Interventions: Other: Masaj
- Control Group (No Intervention): Massage will not be applied to the control group; intervention scales will be applied by taking vital signs after waiting until the massage application in the group (20 minutes in total) and the rest period (30 minutes).

INTERVENTIONS:
Other: Masaj — Appropriate position is given to the patients. Thumb and finger movements, patting, rubbing and squeezing techniques are used in foot massage. During training, the active hand applies pressure, while the passive hand uses both hands to support the foot. The intervention begins with rubbing and warming the feet. The duration of the foot warming process is approximately 5 minutes, and after the foot warming maneuvers, the methods of moving the thumbs of both hands towards the soles of the feet and spinning the laundry are used. The inner and outer parts of the foot are patted in a balanced way. This caressing movement on both feet is done with these movements in a light and rhythmic way and the massage is completed. Data will be obtained with Patient Descriptive Information Form, Vital Signs Follow-up Form, Surgical Anxiety Scale for Adult Patients, Perianesthesia Comfort Scale, Numerical Pain Scale.
  Arms: Massage Group

SUMMARY:
Aim and objectives:The aim of this study is to examine the effect of foot massage on reducing pain and anxiety and increasing the comfort level in patients undergoing laparoscopic cholecystectomy.

Design:The study is a randomized controlled experimental study with a pretest posttest control group.

Methods:This study will be carried out in Niğde Ömer Halisdemir University Training and Research Hospital General Surgery Clinic. Participants were divided into massage group and control group. Vital signs of the massage group will be taken 2 hours before the operation and Surgical Anxiety Scale will be applied to adult patients (n=40). At this stage, the patient's both feet will be massaged for a total of 20 minutes, 10 minutes each. Vital signs and anxiety status of the patients will be evaluated 30 minutes after the procedure. Postoperative vital signs, pain severity, anxiety and comfort level will be evaluated and after the evaluation, a foot massage will be applied to both feet of the patient for 10 minutes, for a total of 20 minutes. Vital signs and pain levels of the patients will be evaluated at the 5th, 30th, 60th, 90th and 120th minutes after the massage, and their comfort and anxiety levels will be evaluated at the 30th minute. The same data will be collected from patients in the control group (n=40) without foot massage. Data will be collected from Patient Descriptive Information Form, Vital Signs Follow-up Form, Surgical Anxiety Scale for Adult Patients, Perianesthesia Comfort Scale, Numerical Pain Scale.will be used.

DETAILED DESCRIPTION:
The study is a randomized controlled experimental study with pre-test post-test control group.The independent variable of the study is foot massage application, the dependent variables are preoperative anxiety level, postoperative pain severity, vital signs (blood pressure, pulse, number of breaths, body temperature, oxygen saturation), anxiety level and comfort level.The research will be conducted at the General Surgery Clinic of Niğde Ömer Halisdemir University Training and Research Hospital.Patients admitted to the General Surgery Clinic for Laparocopic Cholecystectomy surgery after being admitted to the service: The anamnesis form is filled out, the file containing the examinations is prepared,the hunger condition is questioned, the necessary preparations are made for the patient to go to the surgery and the transfer to the operating room is ensured. After the operation; vital signs are checked in postoperative care. The treatment protocol steps are applied in the clinic. Within these steps: I . Usually 2000cc mayi is prepared (LR, 5% Dextrose,0.9% NaCl) II. Antibiotics are administered according to the form specified at the doctor's request (Cefazol or Desefin 2 x 1 V.b.). III. Analgesics are applied according to the patient's condition and the patient's prescription (Oxamen, Tilcotil, Dolantin, Dichlorone, Voltaren, Novalgine) A power analysis was performed to determine the number of people to be included in the research. The strength of the test was calculated with the G*Power 3.1 program. Similar references have been made in the relevant literature. According to the mean and standard deviation values of the Perianesthesia Comfort Scale (PCS) and Numerical Pain Scale (NPS) of the study, the sample size was calculated as 14 people for PPE values and 76 people for PPE values. The study should reach 76 people, including 38 people for each group at the 95% power, 5% significance level and 0.768 effect size. Considering the decrease in the number of patients, it is aimed to recruit a total of 80 people, 40 for each group, to the study.

It was taken by randomization according to the order of arrival in order to avoid bias in the people who will be included in the study.Randomization table "https://www.random.org " it was created using the address. To Investigate the received subjects were matched with the randomization table according to the order of arrival and divided into groups impartially.

Criteria for Inclusion in the Research:

* Who volunteered to participate in the study,

  * who is 18 years of age or older,
  * Without communication difficulties and mental disabilities related to vision, hearing and speech,
  * The hypertension problem has been brought under control,
  * Blood pressure measurement does not need to be performed on an outpatient basis,
  * Any complications after surgery (bleeding, nausea, vomiting, etc.) that did not occur,
* Performing cholecystectomy surgery,

  * Having a pain assessment score of 4 and above after surgical intervention,
  * For patients in the experimental group; infectious disease, local infection, open lesion/wound, scar tissue, edema on the skin,hematoma, thrombophlebitis, deep vein thrombosis, lymphangitis, coagulation disorder, varicose veins, osteoporosis, osteomyelitis.

Exclusion Criteria:

After the surgical procedure, severe bleeding, nausea, vomiting, such as any developing complications,

* Patient-controlled analgesia (HKA) is applied for pain control after surgical intervention
* Patients who have at least one drain placed at the surgery site are excluded from the sample, as it may affect the pain level will be released hepatitis, inflammatory and degenerative joint diseases, advanced neuropathy due to diabetes, in the toes who has not experienced deformity, recent fracture, dislocation, rupture of November muscle fiber, tendon or fascia,
* No analgesic applied before the first attempt planned to be applied after surgery,

  • Any medicine, etc. non-substance abuse,
* No chronic pain in any area of the body, • All patients who are not pregnant will be included in the scope of the sample

Termination Criteria:

During the application, the individual feels uncomfortable or leaves the study the work will be terminated if requested.

Data Collection Tools:

A two-part Patient Identification Information Form, Life Findings, Follow-up Form, Surgical Anxiety Scale for Adult Patients, Perianesthesia Comfort Scale, and Numerical Pain Scale will be used to collect the data.

Introductory Patient Information Form:

I of this form prepared by the researcher in accordance with the relevant literature.In the section; age, gender, height, weight, educational level, marital status, occupation, smoking and alcohol use and methods of coping with pain, II. In the section, there are questions that question situations such as the location, nature of pain, the use of analgesics.

Collection of Data:

The subjects included in the study were matched with the randomization table according to the order of arrival and divided into intervention and control groups impartially. From these separated groups, the intervention group will be given routine clinical treatment and standard nursing care, as well as foot massage, while the control group will not be given any treatment, routine clinical treatment and standard nursing care will be provided.

Applications to be Made to the Intervention Group:

Foot massage applied to intervention group patients is about this it will be carried out in accordance with the information received in the course by the researcher who has received training and has a certificate.

Vaseline or liquid glycerin recommended by the massage instructor to facilitate hand movements during massage it will be made using. Information about the procedure to patients who meet the criteria for admission to the study on the day of the operation oral and written permissions will be obtained using the Informed Voluntary Consent form. Patient Information Form the scales will be filled in and introduced. Routine treatment applied to the intervention group in the clinic before and after surgery,standard nursing care and foot massage; will be applied. The intervention group's vital signs 2 hours before surgery the findings will be taken and the Surgical Anxiety Scale For Adult Patients will be applied to this group. From the scale evaluation then, foot massage will be applied to each foot for a total of 20 minutes, including 10 minutes.

Vital signs will be taken 30 minutes after the massage application is completed and the anxiety level will be evaluated with the Surgical Anxiety Scale for Adult Patients. The application of postoperative scales and foot massage will be performed 3 hours after the operation, the patients' vital signs will be taken and the pain severity will be evaluated with a Numerical Pain Scale. Simultaneously, the patients' comfort will be evaluated using the Perianesthesia Comfort Level Scale and their anxiety levels will be evaluated using the Surgical Anxiety Scale. After the evaluation, foot massage will be performed on each foot for a total of 20 minutes from 10 minutes. Foot massage will be applied to patients with a pain severity score of 4 and above. After the massage, taking into account the literature information, 5., 30., 60., 90. and 120. the severity of pain in minutes and vital signs it will be evaluated. Anxiety and comfort levels are 30. it will be evaluated per minute. Analgesics applied during discharge and usage amounts will be recorded.

Intervention Group Massage Protocol:

The neck, waist and knee parts of the patients are supported and the semi-fowler or supine position is given to the patients in bed.

* It is necessary for the practitioner to bring the hands to the appropriate temperature by washing them and to apply with short nails.
* The practitioner passes to the patient's feet, bringing the patient's feet to the chest level of the person applying the position is given and eye contact is made with the patient during the application.
* Thumb and finger movements, stroking, rubbing and squeezing movements technique in foot massage application is used. During the adjustment of the pressure intensity, the physical structure of the person, age, etc. characteristics are taken into account. Deep, strong and slow pressure movements in order to relieve and relieve pain, light, fast, progressive pressure movements are stimulating it is applied for the purpose of being. During the application, the active hand applies pressure and the passive hand uses two hands to support the foot the hand is used at the same time.
* The intervention begins by rubbing and warming the feet. After the heating process, first of all, more than one application.it starts with the right foot, which has a nerve end zone and sensitivity, then moves to the left foot.
* The foot heating process time is about 5 minutes, and the foot heating process maneuvers are called "Achilles tendon stretching, wrist relaxation, walking the thumbs of both hands on the sole of the foot and laundry tightening methods are used".
* The pituitary gland and hypothalamus reflex points on the big toe are massaged with caterpillar movement. The same process it is also applied to the other fingers respectively.
* In the form of a worm walk with thumbs from top to bottom and from bottom to top to spinal cord reflex points massage is performed.
* Massage is performed on the intestinal reflex point and adrenal glands reflex points for approximately 3 minutes.
* To the solar plexus area (sympathetic neural networks in the abdominal cavity area to send a warning to the entire body the biggest one) is massaged. Stay in this area by applying a light pressure massage for about 2-3 minutes.
* The inner and outer parts of the foot are patted in a balancing manner. This patting movement on both feet in a light and rhythmic way it is applied and the massage is finished with these movements

Applications to be Made to the Control Group:

The control group that meets the criteria for admission to the study will be informed about the procedure before the surgery on the day of the surgery and oral and written permissions of this group will be obtained using the Informed Voluntary Consent form. The scales will be introduced by filling out the Patient Information Form. The control group vital signs will be taken 2 hours before the operation and Surgical Anxiety Scale For Adult Patients in this group will be applied. No massage application will be performed after the scale evaluation; intervention after waiting until the massage application in the group (a total of 20 minutes) and the rest period (30 minutes), vital the findings will be taken again and the anxiety level will be evaluated with the Surgical Anxiety Scale for Adult Patients. When the patient expresses that he has pain after surgery, the Numerical Pain Scale and the severity of pain with vital signs, anxiety and the comfort level will be evaluated. Waiting for the duration of foot massage performed to the intervention group; 5., 30., 60., 90. and 120. the severity of pain and vital signs will be evaluated in minutes. 30. anxiety and comfort level per minute it will be evaluated. Analgesics applied during discharge and usage amounts will be recorded

ELIGIBILITY:
Inclusion Criteria:

Who volunteered to participate in the study,

* those who are 18 years of age or older,

  * Without communication difficulties and mental disabilities related to vision, hearing and speech,
  * Hypertension problem has been controlled,
  * Blood pressure measurement does not need to be performed on an outpatient basis,
* Any complications after surgery (bleeding, nausea, vomiting, etc.) that did not occur,

  * Application of cholecystectomy surgery,
  * Having a pain assessment score of 4 and above after surgical intervention,
  * For patients in the experimental group; infectious disease on the skin, local infection, open lesion/wound, scar tissue, edema,hematoma, thrombophlebitis, deep vein thrombosis, lymphangitis, coagulation disorder, varicose veins, osteoporosis, osteomyelitis, hepatitis, inflammatory and degenerative joint diseases, advanced neuropathy due to diabetes, on the toes deformity, November, who has not recently experienced fractures, dislocations, ruptures of muscle fibers, tendons or fascia,
  * Analgesic is not applied before the first attempt, which is planned to be applied after the operation,
* Any medication, etc. without substance abuse,

  * No chronic pain in any part of the body,
* All patients who are not pregnant will be included in the sample.

Exclusion Criteria:

Any complications such as severe bleeding, nausea, vomiting develop after surgical intervention.,

* Patient-controlled analgesia (HKA) is applied for pain control after surgical intervention
* Patients who have at least one drain placed at the surgical site are excluded from the sample, as this may affect the level of pain he will be released.

Termination Criteria: The individual feels uncomfortable during the application or to leave the study if he wants, the work will be terminated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Perianesthesia Comfort Scale | Two days
  PCS consisting of 24 items and before the individual's surgery, it is a 6-point Likert-type scale that questions their general thoughts and feelings about the process during and after. The scale scoring varies between 1 and 6 points Dec, the scale questions are scored as 1= "I Strongly Disagree" 6= "I Strongly Agree".The highest total score of PCS is 144 and the lowest total score is 24.

SECONDARY OUTCOMES:
Numerical Pain Scale | Two days
  This scale, which aims to determine the severity of pain, aims to explain the patient's pain with numbers. It starts with the absence of pain on numerical scales (0) and reaches up to the level of unbearable pain (10).It is preferred due to the fact that it is an understandable and easily applied scale used by researchers at international and national levels to facilitate the identification of patients' pain severity, facilitate scoring and reduce pain.

OTHER OUTCOMES:
Surgical Anxiety Scale for Adult Patients | Two days
  The scale has been prepared in order to determine the surgical anxiety levels of the sick individuals who will undergo surgical operation.The sub-dimensions of the scale are health-related concerns (7., 9., 10., 11., 12. and 13. substances),concerns about recovery time(14., 15., 16. and 17. substances) and concerns about the surgical procedure (1., 2., 4. and 8. substances) and concerns about invasive procedures (3., 5. and 6. there are 4 of them (substances).The scale items are scored as 0 = "I am not worried at all", 1 = "I am very little worried", 2 = "I am partially worried", 3 = "I am very worried" and 4 = "I am extremely worried".The lowest score that can be taken from the scale is 0, the highest score is 68.

CONTACTS AND LOCATIONS:
Locations (1):
- Nesibe Sultan ÇINAROĞLU, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No